CLINICAL TRIAL: NCT00289913
Title: An Open, Randomized, Multicenter Study of the Safety, Tolerability, and Immunogenicity of VAQTA™ Given Concomitantly With PedvaxHIB™ and Infanrix™ in Healthy Children 15 Months of Age
Brief Title: Concomitant Use of Hepatitis A Vaccine, Inactivated With Haemophilus b Conjugate Vaccine (Meningococcal Protein Conjugate) and Diphtheria and Tetanus Toxoids and Acellular Pertussis Vaccine Adsorbed Given to Healthy Children 15 Months of Age (V251-068)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V251-068; 2005_076
Record Dates: First submitted 2006-02-08; First posted 2006-02-10 (Estimated); Results first posted 2011-07-07 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis A Virus
Keywords: Hepatitis A virus
MeSH Terms: conditions — Hepatitis

ARMS (5):
- VAQTA™, PedvaxHIB™ and Infanrix™/VAQTA™ (Stage 1) (Experimental): Day 1: VAQTA™ (first dose), PedvaxHIB™ and Infanrix™ were administered concomitantly at different injection sites.
  Week 24: The second dose of VAQTA™ was administered.
  Interventions: Biological: Comparator: VAQTA™; Biological: Comparator: Infanrix™; Biological: Comparator: PedvaxHIB™
- PedvaxHIB™ and Infanrix™/VAQTA™/VAQTA™ (Stage 1) (Experimental): Day 1: PedvaxHIB™ and Infanrix™ were administered concomitantly at different injection sites.
  Week 4: The first dose of VAQTA™ was administered.
  Week 28: The second dose of VAQTA™ was administered.
  Interventions: Biological: Comparator: VAQTA™; Biological: Comparator: Infanrix™; Biological: Comparator: PedvaxHIB™
- VAQTA™, PedvaxHIB™/VAQTA™ (Stage 1) (Experimental): Day 1: VAQTA™ (first dose) and PedvaxHIB™ were administered concomitantly at different injection sites.
  Week 24: The second dose of VAQTA™ was administered.
  Interventions: Biological: Comparator: VAQTA™; Biological: Comparator: PedvaxHIB™
- PedvaxHIB™/VAQTA™/VAQTA™ (Stage 1) (Experimental): Day 1: PedvaxHIB™ was administered.
  Week 4: The first dose of VAQTA™ was administered.
  Week 28: The second dose of VAQTA™ was administered.
  Interventions: Biological: Comparator: VAQTA™; Biological: Comparator: PedvaxHIB™
- VAQTA™/VAQTA™ (Stage 2) (Experimental): Day 1: The first dose of VAQTA™ was administered.
  Week 24: The second dose of VAQTA™ was administered.
  Interventions: Biological: Comparator: VAQTA™

INTERVENTIONS:
Biological: Comparator: VAQTA™ — VAQTA™ (Hepatitis A Vaccine, Inactivated).
  Two intramuscular 0.5-mL doses of VAQTA™ were administered 24 weeks apart, with the second dose being administered prior to 24 months of age.
Biological: Comparator: Infanrix™ — Infanrix™ (Diphtheria and Tetanus Toxoids and Acellular Pertussis
  Vaccine Adsorbed, GlaxoSmithKline).
  One intramuscular 0.5-mL injection of Infanrix™ was administered at the first study visit.
  Arms: PedvaxHIB™ and Infanrix™/VAQTA™/VAQTA™ (Stage 1); VAQTA™, PedvaxHIB™ and Infanrix™/VAQTA™ (Stage 1)
Biological: Comparator: PedvaxHIB™ — PedvaxHIB™ (Haemophilus B Conjugate Vaccine [Meningococcal Protein Conjugate]).
  One intramuscular 0.5-mL injection of PedvaxHIB™ was administered at the first study visit.
  Other Names: One intramuscular 0.5-mL injection of PedvaxHIB™ was administered to all subjects at the first study; visit in all treatment groups in the study.
  Arms: PedvaxHIB™ and Infanrix™/VAQTA™/VAQTA™ (Stage 1); PedvaxHIB™/VAQTA™/VAQTA™ (Stage 1); VAQTA™, PedvaxHIB™ and Infanrix™/VAQTA™ (Stage 1); VAQTA™, PedvaxHIB™/VAQTA™ (Stage 1)

SUMMARY:
This two-stage study evaluates the immunogenicity, safety, and tolerability of the administration of VAQTA™ (Hepatitis A Vaccine, Inactivated) concomitantly with PedvaxHIB™ (Haemophilus B Conjugate Vaccine [Meningococcal Protein Conjugate]) and Infanrix™ (Diphtheria and Tetanus Toxoids and Acellular Pertussis Vaccine Adsorbed, GlaxoSmithKline) versus the administration of VAQTA™ in healthy children 15 months of age at study entry.

DETAILED DESCRIPTION:
In stage I, VAQTA™ given concomitantly with Infanrix™ and/or PedvaxHIB™ was evaluated.

In stage 2: Two (2) doses of the VAQTA™ vaccine were administered at least 6 months apart. Safety data was collected after each dose.

ELIGIBILITY:
Inclusion Criteria:

* Stage 1) Healthy males and females 15 months of age with no active liver disease and a negative history of hepatitis A who have been vaccinated against Haemophilus influenzae type b (Hib), diphtheria, tetanus, and pertussis diseases
* Stage 2) Healthy males and females 12 to 17 months of age with no active liver disease and a negative history of hepatitis A

Exclusion Criteria:

* Stage 1) Males and females previously vaccinated with hepatitis A vaccine, any immune deficiency, a history of allergy to any of the vaccine components, a history of seizure disorder or a neurologic disorder that would contraindicate pertussis vaccine, or a bleeding disorder
* Stage 2) Males and females previously vaccinated with hepatitis A vaccine, any immune deficiency, a history of allergy to any of the vaccine components, or a history of bleeding disorder

Ages: 12 Months to 17 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1274 (Actual)
Dates: Start 2006-04; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Petrecz M, Ramsey KP, Stek JE, Martin JC, Klopfer SO, Kuter B, Schodel FP, Lee AW. Concomitant use of VAQTA with PedvaxHIB and Infanrix in 12 to 17 month old children. Hum Vaccin Immunother. 2016;12(2):503-11. doi: 10.1080/21645515.2015.1080395. PMID 26308112

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In Stage I, a total of 620 participants were randomized to receive study vaccinations. However for 3 participants, the Health Insurance Portability and Accountability Act (HIPAA) and/or Informed Consent Form was not signed by the parents in error. Therefore a total of 617 participants were included in Stage I. 654 participants started Stage II.
Pre-assignment Details: For this study: Visit 1 was on Day 1 (for Stage I and Stage II). Visit 2 was at Week 4 (Stage I) and Week 2 (Stage II). Visit 3 was at Week 24/Week 28 (Stage I) and Week 24 (Stage II). Visit 4 was at Week 28/Week 32 (Stage I) and Week 26 (Stage II). For safety, participants were followed for 14 days after each vaccination (safety follow-up [F/U]).
Groups:
- VAQTA™, PedvaxHIB™ and Infanrix™/ VAQTA™ (Stage 1): Day 1: VAQTA™ (first dose), PedvaxHIB™ and Infanrix™ were administered concomitantly at different injection sites.
  Week 24: The second dose of VAQTA™ was administered.
- PedvaxHIB™ and Infanrix™/ VAQTA™/ VAQTA™ (Stage 1): Day 1: PedvaxHIB™ and Infanrix™ were administered concomitantly at different injection sites.
  Week 4: The first dose of VAQTA™ was administered.
  Week 28: The second dose of VAQTA™ was administered.
- VAQTA™, PedvaxHIB™/ VAQTA™ (Stage 1): Day 1: VAQTA™ (first dose) and PedvaxHIB™ were administered concomitantly at different injection sites.
  Week 24: The second dose of VAQTA™ was administered.
- PedvaxHIB™/ VAQTA™/ VAQTA™ (Stage 1): Day 1: PedvaxHIB™ was administered.
  Week 4: The first dose of VAQTA™ was administered.
  Week 28: The second dose of VAQTA™ was administered.
- VAQTA™/ VAQTA™ (Stage 2): Day 1: The first dose of VAQTA™ was administered.
  Week 24: The second dose of VAQTA™ was administered.
Period: Visit 1 (Stage I and Stage II)
Arm/Group | VAQTA™, PedvaxHIB™ and Infanrix™/ VAQTA™ (Stage 1) | PedvaxHIB™ and Infanrix™/ VAQTA™/ VAQTA™ (Stage 1) | VAQTA™, PedvaxHIB™/ VAQTA™ (Stage 1) | PedvaxHIB™/ VAQTA™/ VAQTA™ (Stage 1) | VAQTA™/ VAQTA™ (Stage 2)
Started | 155 | 151 | 159 | 152 | 654 (Participants were enrolled during Stage II.)
Completed | 146 | 135 | 150 | 141 | 645
Not Completed | 9 | 16 | 9 | 11 | 9
Not completed — Protocol deviation during safety F/U | 0 | 1 | 0 | 0 | 0
Not completed — Lost during safety F/U | 3 | 2 | 2 | 2 | 1
Not completed — Withdrew consent during safety F/U | 2 | 2 | 0 | 2 | 2
Not completed — Moved during safety F/U | 0 | 0 | 0 | 0 | 1
Not completed — Other reasons during safety F/U | 0 | 0 | 0 | 1 | 0
Not completed — Protocol deviation after safety F/U | 1 | 2 | 0 | 0 | 0
Not completed — Lost after safety F/U | 2 | 1 | 0 | 0 | 5
Not completed — Withdrew consent after safety F/U] | 0 | 8 | 5 | 6 | 0
Not completed — Other reasons after safety F/U | 1 | 0 | 2 | 0 | 0
Period: Visit 2 (Stage I and Stage II)
Arm/Group | VAQTA™, PedvaxHIB™ and Infanrix™/ VAQTA™ (Stage 1) | PedvaxHIB™ and Infanrix™/ VAQTA™/ VAQTA™ (Stage 1) | VAQTA™, PedvaxHIB™/ VAQTA™ (Stage 1) | PedvaxHIB™/ VAQTA™/ VAQTA™ (Stage 1) | VAQTA™/ VAQTA™ (Stage 2)
Started | 146 | 135 | 150 | 141 | 645 (No vaccine administered at Visit 2 (Stage II), therefore there was no safety F/U period.)
Completed | 131 | 114 | 140 | 135 | 605
Not Completed | 15 | 21 | 10 | 6 | 40
Not completed — Protocol deviation during safety F/U | 0 | 0 | 1 | 0 | 0
Not completed — Lost during safety F/U | 8 | 11 | 2 | 2 | 0
Not completed — Subject moved during safety F/U | 0 | 1 | 0 | 0 | 0
Not completed — Withdrew consent during safety F/U | 3 | 2 | 1 | 0 | 0
Not completed — Other reasons during safety F/U | 1 | 0 | 1 | 0 | 0
Not completed — Protocol deviation after safety F/U | 0 | 1 | 3 | 1 | 0
Not completed — Lost after safety F/U | 2 | 5 | 0 | 3 | 0
Not completed — Withdrew consent after safety F/U | 0 | 1 | 2 | 0 | 0
Not completed — Other reasons after safety F/U] | 1 | 0 | 0 | 0 | 0
Not completed — Protocol deviation (Stage II) | 0 | 0 | 0 | 0 | 7
Not completed — Lost (Stage II) | 0 | 0 | 0 | 0 | 11
Not completed — Moved (Stage II) | 0 | 0 | 0 | 0 | 6
Not completed — Withdrew consent (Stage II) | 0 | 0 | 0 | 0 | 7
Not completed — Other reasons (Stage II) | 0 | 0 | 0 | 0 | 9
Period: Visit 3 (Stage I and Stage II)
Arm/Group | VAQTA™, PedvaxHIB™ and Infanrix™/ VAQTA™ (Stage 1) | PedvaxHIB™ and Infanrix™/ VAQTA™/ VAQTA™ (Stage 1) | VAQTA™, PedvaxHIB™/ VAQTA™ (Stage 1) | PedvaxHIB™/ VAQTA™/ VAQTA™ (Stage 1) | VAQTA™/ VAQTA™ (Stage 2)
Started | 131 | 114 | 140 | 135 | 605
Completed | 122 | 106 | 138 | 131 | 597
Not Completed | 9 | 8 | 2 | 4 | 8
Not completed — Protocol deviation during safety F/U | 0 | 1 | 0 | 0 | 0
Not completed — Lost during safety F/U | 8 | 3 | 1 | 2 | 2
Not completed — Withdrew consent during safety F/U | 0 | 0 | 0 | 1 | 0
Not completed — Other reasons during safety F/U | 0 | 0 | 0 | 0 | 1
Not completed — Lost after safety F/U | 1 | 2 | 0 | 1 | 4
Not completed — Withdrew consent after safety F/U] | 0 | 1 | 1 | 0 | 0
Not completed — Moved after safety F/U | 0 | 0 | 0 | 0 | 1
Not completed — Other reasons after safety F/U | 0 | 1 | 0 | 0 | 0
Period: Visit 4 (Stage I and Stage II)
Arm/Group | VAQTA™, PedvaxHIB™ and Infanrix™/ VAQTA™ (Stage 1) | PedvaxHIB™ and Infanrix™/ VAQTA™/ VAQTA™ (Stage 1) | VAQTA™, PedvaxHIB™/ VAQTA™ (Stage 1) | PedvaxHIB™/ VAQTA™/ VAQTA™ (Stage 1) | VAQTA™/ VAQTA™ (Stage 2)
Started | 122 | 106 | 138 | 131 | 597
Completed | 122 | 106 | 138 | 131 | 597
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VAQTA™, PedvaxHIB™ and Infanrix™/ VAQTA™ (Stage 1) | PedvaxHIB™ and Infanrix™/ VAQTA™/ VAQTA™ (Stage 1) | VAQTA™, PedvaxHIB™/ VAQTA™ (Stage 1) | PedvaxHIB™/ VAQTA™/ VAQTA™ (Stage 1) | VAQTA™/ VAQTA™ (Stage 2) | Total
Number analyzed (Participants) | 155 | 151 | 159 | 152 | 654 | 1271
Age, Customized [Number; unit: participants] — Months between the birthdate and consent date.
  participants
    Between 12 and 18 months | 155 | 151 | 159 | 152 | 654 | 1271
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 67 | 70 | 73 | 319 | 603
  Male | 81 | 84 | 89 | 79 | 335 | 668

OUTCOME MEASURES:

1. Primary Outcome: Seropositivity Rate (SPR) to Hepatitis A
Description: SPR is the percent of participants with Hepatitis A antibody titers >= 10 milli-International Units/milliliter (mIU/mL), 4 weeks after dose 2 of VAQTA™ regardless of their initial serostatus. Antibody titers to Hepatitis A virus (HAV) were detected in participants' serum samples using an Enzyme Immunoassay (EIA).
Time Frame: 4 weeks after dose 2 of VAQTA™
Population: The per-protocol population, which consisted of all Stage I participants who received vaccinations within the specified day ranges, completed appropriate follow-up, and were without any pre-specified protocol violations.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | VAQTA™, PedvaxHIB™ and Infanrix™/ VAQTA™ (Stage 1) | PedvaxHIB™ and Infanrix™/ VAQTA™/ VAQTA™ (Stage 1) | VAQTA™, PedvaxHIB™/ VAQTA™ (Stage 1) | PedvaxHIB™/ VAQTA™/ VAQTA™ (Stage 1) | VAQTA™/ VAQTA™ (Stage 2)
Number analyzed (Participants) | 94 | 78 | 114 | 105 | 0
Percentage of participants | 100 [96.2 to 100] | 100 [95.4 to 100] | 100 [96.8 to 100] | 100 [96.5 to 100] |

2. Primary Outcome: Antibody Response Rate to Haemophilus Influenzae Type b (Hib)
Description: Antibodies to the Hib capsular polysaccharide (polyribosylribitol phosphate [PRP]) are assessed in participants serum using radioimmunoassay (RIA). The limit of detection (LOD) for the RIA is 6.60 ng/mL.
  The antibody response rate is defined as the percentage of participants with anti-PRP titers >1.0 mcg/mL, 4 weeks postvaccination with PedvaxHIB™.
Time Frame: 4 weeks postvaccination with PedvaxHIB™
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | VAQTA™, PedvaxHIB™ and Infanrix™/ VAQTA™ (Stage 1) | PedvaxHIB™ and Infanrix™/ VAQTA™/ VAQTA™ (Stage 1) | VAQTA™, PedvaxHIB™/ VAQTA™ (Stage 1) | PedvaxHIB™/ VAQTA™/ VAQTA™ (Stage 1) | VAQTA™/ VAQTA™ (Stage 2)
Number analyzed (Participants) | 106 | 99 | 110 | 109 | 0
Percentage of participants | 98.1 [93.4 to 99.8] | 97.0 [91.4 to 99.4] | 97.3 [92.2 to 99.4] | 97.2 [92.2 to 99.4] |

3. Primary Outcome: Number of Participants With Adverse Events (AE)
Description: Systemic and injection site AEs were collected from participants receiving
  * VAQTA™ concomitantly with Infanrix™ and PedvaxHIB™ or PedvaxHIB™ (Stage I)
  * VAQTA™ non-concomitantly with Infanrix™ and PedvaxHIB™ or PedvaxHIB™ (Stage I)
  * VAQTA™ administered alone (Stage II)
  Safety data was collected on a standardized Vaccination Report Card (VRC)
  following each dose. Participants returned the VRC after the safety follow-up period for each dose of VAQTA™. AEs determined by the investigator to be possibly, probably or definitely related to the vaccine are reported as Vaccine-related AE.
Time Frame: Days 1 to 14 after any dose of VAQTA™ for systemic AEs, and Days 1 to 5 after any dose of VAQTA™ for injection-site AEs
Population: Participants administered at least one dose of vaccine, for whom follow-up was available.
Measure: Number; unit: Participants
Groups:
- Concomitant VAQTA™ With Infanrix™ and PedvaxHIB™ or PedvaxHIB™: All participants receiving VAQTA™ Concomitantly with Infanrix™ and PedvaxHIB™ or PedvaxHIB™ were pooled for safety analysis; and includes participants from Groups 1: VAQTA™, PedvaxHIB™ and Infanrix™/VAQTA™ (Stage 1); and Group 3: VAQTA™, PedvaxHIB™/VAQTA™ (Stage 1).
- Non-concomitant VAQTA™ Separate From Infanrix™ and PedvaxHIB™: All participants receiving VAQTA™ non-concomitantly with Infanrix™ and PedvaxHIB™ or PedvaxHIB™ were pooled for safety analysis; and includes participants from Groups 2: PedvaxHIB™ and Infanrix™/VAQTA™/VAQTA™ (Stage 1); and Group 4: PedvaxHIB™/VAQTA™/VAQTA™ (Stage 1).
- VAQTA™/VAQTA™: All participants receiving VAQTA™ alone (from Stage II) on Day 1 and Day 24.
Arm/Group | Concomitant VAQTA™ With Infanrix™ and PedvaxHIB™ or PedvaxHIB™ | Non-concomitant VAQTA™ Separate From Infanrix™ and PedvaxHIB™ | VAQTA™/VAQTA™
Number analyzed (Participants) | 302 | 256 | 647
Participants
  With no AE | 63 | 86 | 181
  With one or more AE | 239 | 170 | 466
  ---injection-site AE | 167 | 116 | 249
  ---sytemic AE | 183 | 119 | 395
  With vaccine-related (VR) AE | 192 | 129 | 328
  ---injection-site AE (VR) | 164 | 116 | 249
  ---sytemic AE (VR) | 91 | 42 | 147
  With serious AE | 0 | 1 | 2
  With serious AE (VR) | 0 | 0 | 0
  Who died | 0 | 0 | 0
  Who discontinued due to AE | 0 | 0 | 0
  Who discontinued due to serious AE | 0 | 0 | 0

4. Primary Outcome: Geometric Mean Titers (GMTs) to Antibodies for the Pertussis Toxin (PT), Pertussis Filamentous Hemagglutinin Antibody (FHA), and Pertactin (PRN) Components of Infanrix™
Description: GMTs for antibodies to PT, FHA, and PRN were measured in serum samples of participants vaccinated with Infanrix™.
  IgG antibodies to PT were assessed using the anti-pertussis toxin enzyme-linked immunosorbent assay (anti-PT ELISA), with the LOD of 2.4 ELU/mL.
  IgG antibodies to FHA were assessed using the anti-pertussis filamentous hemagglutinin enzyme-linked immunosorbent assay (anti-FHA ELISA), with the LOD of 2.0 ELU/mL.
  IgG antibodies to PRN were assessed using the anti-pertussis pertactin enzyme-linked immunosorbent assay (anti-PRN ELISA), with the LOD of 3.3 ELU/mL.
Time Frame: 4 weeks postvaccination with Infanrix™
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA units per mL (ELU/mL)
Arm/Group | VAQTA™, PedvaxHIB™ and Infanrix™/ VAQTA™ (Stage 1) | PedvaxHIB™ and Infanrix™/ VAQTA™/ VAQTA™ (Stage 1) | VAQTA™, PedvaxHIB™/ VAQTA™ (Stage 1) | PedvaxHIB™/ VAQTA™/ VAQTA™ (Stage 1) | VAQTA™/ VAQTA™ (Stage 2)
Number analyzed (Participants) | 85 | 83 | 0 | 0 | 0
ELISA units per mL (ELU/mL)
  Pertussis PT | 69.2 [57.4 to 83.5] | 51.7 [41.5 to 64.5] |  |  |
  Pertussis FHA | 253.8 [215.3 to 299.2] | 249.2 [200.6 to 309.5] |  |  |
  PRN | 333.5 [267.3 to 416.1] | 358.5 [282.7 to 454.7] |  |  |

ADVERSE EVENTS:
Groups:
- PedvaxHIB™/ VAQTA™/ VAQTA™ (Stage I): Day 1: PedvaxHIB™ was administered.
  Week 4: The first dose of VAQTA™ was administered.
  Week 28: The second dose of VAQTA™ was administered.
Arm/Group | VAQTA™, PedvaxHIB™ and Infanrix™/ VAQTA™ (Stage 1) | PedvaxHIB™ and Infanrix™/ VAQTA™/ VAQTA™ (Stage 1) | VAQTA™, PedvaxHIB™/ VAQTA™ (Stage 1) | PedvaxHIB™/ VAQTA™/ VAQTA™ (Stage I) | VAQTA™/ VAQTA™ (Stage 2)
Serious Adverse Events (participants affected / at risk) | 0/150 | 2/145 | 0/152 | 2/146 | 2/641
Other Adverse Events (participants affected / at risk) | 116/150 | 74/145 | 123/152 | 88/146 | 426/641
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VAQTA™, PedvaxHIB™ and Infanrix™/ VAQTA™ (Stage 1) (N=150) | PedvaxHIB™ and Infanrix™/ VAQTA™/ VAQTA™ (Stage 1) (N=145) | VAQTA™, PedvaxHIB™/ VAQTA™ (Stage 1) (N=152) | PedvaxHIB™/ VAQTA™/ VAQTA™ (Stage I) (N=146) | VAQTA™/ VAQTA™ (Stage 2) (N=641)
LYMPHADENITIS (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTITIS MEDIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SUBCUTANEOUS ABSCESS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FOREIGN BODY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VAQTA™, PedvaxHIB™ and Infanrix™/ VAQTA™ (Stage 1) (N=150) | PedvaxHIB™ and Infanrix™/ VAQTA™/ VAQTA™ (Stage 1) (N=145) | VAQTA™, PedvaxHIB™/ VAQTA™ (Stage 1) (N=152) | PedvaxHIB™/ VAQTA™/ VAQTA™ (Stage I) (N=146) | VAQTA™/ VAQTA™ (Stage 2) (N=641)
DIARRHOEA (Gastrointestinal disorders) | 21 (23) | 8 (10) | 16 (17) | 8 (10) | 50 (54)
TEETHING (Gastrointestinal disorders) | 3 (3) | 3 (4) | 8 (8) | 9 (9) | 56 (69)
VOMITING (Gastrointestinal disorders) | 7 (7) | 4 (4) | 10 (11) | 8 (8) | 27 (31)
INJECTION SITE ERYTHEMA (General disorders) | 48 (62) | 30 (39) | 42 (55) | 43 (58) | 139 (174)
INJECTION SITE PAIN (General disorders) | 75 (98) | 40 (54) | 62 (83) | 55 (71) | 203 (264)
INJECTION SITE SWELLING (General disorders) | 36 (42) | 15 (19) | 26 (30) | 26 (30) | 73 (88)
IRRITABILITY (General disorders) | 28 (35) | 13 (13) | 13 (13) | 11 (14) | 79 (102)
PYREXIA (General disorders) | 43 (58) | 24 (28) | 42 (47) | 23 (24) | 106 (123)
NASOPHARYNGITIS (Infections and infestations) | 21 (22) | 8 (8) | 7 (9) | 4 (4) | 19 (19)
OTITIS MEDIA (Infections and infestations) | 9 (9) | 4 (5) | 19 (19) | 9 (10) | 38 (39)
RHINITIS (Infections and infestations) | 11 (13) | 1 (2) | 5 (5) | 0 (0) | 10 (12)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 9 (9) | 5 (6) | 23 (25) | 8 (10) | 65 (69)
COUGH (Respiratory, thoracic and mediastinal disorders) | 13 (16) | 3 (3) | 12 (12) | 6 (6) | 48 (50)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 11 (13) | 5 (5) | 13 (14) | 6 (10) | 57 (65)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. SPONSOR review can be expedited to meet publication guidelines.